CLINICAL TRIAL: NCT02235532
Title: Effects of Aloe Vera Toothpaste on Periodontal Parameters of Patients With Gingivitis
Brief Title: Effects of Aloe Vera Toothpaste on Periodontal Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Islamic Azad University, Sanandaj (Other)
Responsible Party: Principal Investigator, Ferena Sayar, assistant professor, Islamic Azad University, Sanandaj
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: IRCT2014040517053N2
Record Dates: First submitted 2014-08-30; First posted 2014-09-10 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Gingivitis
Keywords: clinical trial; oral hygiene; Gingivitis; Aloevera; Toothpaste; anti-inflammatory agents
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Foramen Herbal Aloe toothpaste (Experimental): test group was asked to brush the teeth with Foramen Herbal Aloe toothpaste for 30 days once a day.
  Interventions: Other: Foramen Herbal Aloe toothpaste
- use of fluoride toothpaste (signal) (Active Comparator): use of a fluoride toothpaste (signal) in control group once a day for 30 days .
  Interventions: Other: fluoride toothpaste

INTERVENTIONS:
Other: Foramen Herbal Aloe toothpaste — use of aloe-vera toothpaste for 30 days in the test group.
  Arms: Foramen Herbal Aloe toothpaste
Other: fluoride toothpaste — use of signal toothpaste once a day for 30 days in the control group.
  Other Names: signal
  Arms: use of fluoride toothpaste (signal)

SUMMARY:
This study aimed to assess the effects of Aloe Vera toothpaste on dental plaque and gingivitis.

The single-blind cross-over clinical trial was conducted on 20 dental students (10 males and 10 females with a mean age of 24.5±4 yrs.) with gingivitis. Students were randomly divided into 2 groups. The first group used Aloe Vera toothpaste for 30 days. A 2-week wash-out period was allowed and then subjects used fluoride toothpaste for the next 30 days . This order was reversed in group 2.

DETAILED DESCRIPTION:
Toothpastes are used with tooth brushing to better control microbial plaque. Herbal toothpastes have recently gained attention. This study aimed to assess the effects of Aloe Vera toothpaste on dental plaque and gingivitis.

This single-blind cross-over clinical trial was conducted on 20 dental students (10 males and 10 females with a mean age of 24.5±4 yrs.) with gingivitis. Students were randomly divided into 2 groups. The first group used Aloe Vera toothpaste for 30 days and then their plaque index (PI) and gingival index (GI) were recorded. A 2-week wash-out period was allowed and then subjects used fluoride toothpaste for the next 30 days and underwent PI and GI assessment again. This order was reversed in group 2. Wilcoxon-Sign Rank and two way Repeated Measure ANOVA tests were applied for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects were selected among dental students with at least 20 natural teeth without systemic disease
* No periodontal treatment at least 6 months to the study
* No use of systemic antibiotic and anti-inflammatory drugs within the last 3 months, nonsmokers, no pregnancy or lactating women
* Subjects with PD≤3mm, (clinical attachment level)CAL<1mm, PI≥2 and gingival bleeding in more than 30% of the tested areas were enrolled with the diagnosis of plaque-related gingivitis.

Exclusion Criteria:

* Subjects with orthodontic appliances ,multiple bridges, partial denture, multiple caries were excluded from the study

Ages: 20 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-09; Primary Completion 2014-02 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
measuring gingival index | 1-2days
  to compare the efficacy of the aloe-vera toothpaste with a known conventional toothpaste, the gingival index was recorded at baseline and after 30 days of consumption and compared with the two understudy toothpastes.

SECONDARY OUTCOMES:
measuring gingival index | 1-2 days
  to compare the efficacy of the aloe-vera toothpaste with a known conventional toothpaste, the gingival index was recorded at baseline and after 30 days of consumption and compared with the two understudy toothpastes.
measuring plaque index | 1-2 days
  to compare the efficacy of the aloe-vera toothpaste with a known conventional toothpaste, the plaque index was recorded at baseline and after 30 days of consumption and compared with the two understudy toothpastes.

CONTACTS AND LOCATIONS:
Overall Officials: Ferena Sayar, DDS;MSc, Principal Investigator — Tehran Dental Branch, Islamic Azad University,Tehran/Iran
Locations (1):
- Tehran Dental Branch, Islamic azad University, Tehran, Tehran Province, Iran